CLINICAL TRIAL: NCT02168894
Title: A Phase I-II Study of Acupuncture for the Treatment of Chronic, Chemotherapy-Induced Peripheral Neuropathy in Cancer Survivors
Brief Title: SINF: Peripheral Neuropathy in Cancer Survivors
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0930; NCI-2014-01466 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Peripheral Neuropathy
Keywords: Peripheral neuropathy; Chemotherapy-Induced Peripheral Neuropathy; Cancer Survivors; Acupuncture; Electrical stimulation; Nerve function tests; Hand function tests; Balance tests; Questionnaires; Surveys
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Acupuncture Therapy; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 - Acupuncture With Electrical Stimulation (Experimental): Participants in Group 1 have acupuncture sessions with electrical stimulation 3 times a week for 4 weeks, for a total of 12 sessions. Then, take a 2 week break. After that, participant randomly assigned to receive 12 sessions of acupuncture with electrical stimulation as before or not have anymore sessions in this study. Nerve function tests performed at visit before acupuncture and at end of study visit. These tests consist of hand tasks and balance tests. Questionnaires completed at baseline, visit before acupuncture, after 6 and 12 acupuncture visits, and at end of study visit.
  Interventions: Procedure: Acupuncture; Procedure: Nerve Function Tests; Behavioral: Questionnaires
- Group 2 - Acupuncture Sessions Without Electrical Stimulation (Experimental): Participants in Group 2 have acupuncture sessions without electrical stimulation 3 times a week for 4 weeks, for a total of 12 sessions. Then, will take a 2 week break. After that, participant randomly assigned to receive 12 extra sessions of acupuncture without electrical stimulation or not have anymore sessions in this study. Nerve function tests performed at visit before acupuncture and at end of study visit. These tests consist of hand tasks and balance tests. Questionnaires completed at baseline, visit before acupuncture, after 6 and 12 acupuncture visits, and at end of study visit.
  Interventions: Procedure: Acupuncture; Procedure: Nerve Function Tests; Behavioral: Questionnaires
- Group 3 - Waitlist Group (Active Comparator): Participants in Group 3 have acupuncture sessions 3 times per week over 4 weeks for a total of 12 sessions. Participant may or may not have electrical stimulation at these sessions. These sessions will begin 14 weeks after enrollment. Nerve function tests performed at visit before acupuncture and at end of study visit. These tests consist of hand tasks and balance tests. Questionnaires completed at baseline, visit before acupuncture, after 6 and 12 acupuncture visits, and at end of study visit.
  Interventions: Procedure: Acupuncture; Procedure: Nerve Function Tests; Behavioral: Questionnaires

INTERVENTIONS:
Procedure: Acupuncture — Group 1: Acupuncture sessions with electrical stimulation 3 times a week for 4 weeks, for a total of 12 sessions. Then, take a 2 week break. After that, participant randomly assigned to receive 12 sessions of acupuncture with electrical stimulation as before or not have anymore sessions in this study.
  Group 2: Acupuncture sessions without electrical stimulation 3 times a week for 4 weeks, for a total of 12 sessions. Then, will take a 2 week break. After that, participant randomly assigned to receive 12 extra sessions of acupuncture without electrical stimulation or not have anymore sessions in this study.
  Group 3: Acupuncture sessions 3 times per week over 4 weeks for a total of 12 sessions. Participant may or may not have electrical stimulation at these sessions. These sessions will begin 14 weeks after enrollment.
Procedure: Nerve Function Tests — Nerve function tests consisting of hand tasks and balance evaluation performed at visit before acupuncture, and at end of study visit.
Behavioral: Questionnaires — Questionnaire completion at baseline, visit before acupuncture, after 6th and 12th acupuncture session, and at end of study visit.
  Other Names: Surveys

SUMMARY:
The goal of this clinical research study is to learn if one acupuncture treatment approach is more effective than another in helping to relieve neuropathy in cancer patients.

DETAILED DESCRIPTION:
Peripheral neuropathy is a common problem among cancer patients who have received chemotherapy treatment. Acupuncture is a technique that may treat symptoms by inserting very thin, solid, sterile, stainless steel needles into the skin at specific points. Weak electrical stimulation is also applied to the needles to try to improve the treatment effects of the acupuncture.

Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in a roll of dice) to 1 of 3 groups. This is done because no one knows if one study group is better, the same, or worse than the other group.

* If you are in Group 1, you will have will have acupuncture sessions with electrical stimulation 3 times a week for 4 weeks, for a total of 12 sessions. Then, you will take a 2 week break. After that, you will randomly assigned to receive 12 sessions of acupuncture with electrical stimulation as before or not have anymore sessions in this study.
* If you are in Group 2, you will have will have acupuncture sessions without electrical stimulation 3 times a week for 4 weeks, for a total of 12 sessions. Then, you will take a 2 week break. After that, you will randomly assigned to receive 12 extra sessions of acupuncture without electrical stimulation or not have anymore sessions in this study.
* If you are in Group 3, you will have acupuncture sessions 3 times per week over 4 weeks for a total of 12 sessions. You may or may not have electrical stimulation at these sessions. These sessions will begin 14 weeks after you enroll.

Study Visits Before the First Acupuncture Session:

You will return to the clinic about 7-10 days after the screening visit. The following tests will be performed 2 times over a 1-2 week span:

* You will complete 3 questionnaires. The questionnaires will ask about any pain you may be having, about numbness and tingling you may be having, and about other cancer symptoms, such as fatigue and appetite changes. In total, these questionnaires should take 15-20 minutes to complete.
* Your tongue will be checked and you heart rate will be measured. This information will help the study doctor/acupuncturist learn how your body's organs are functioning together.
* If you can become pregnant, urine will be collected for a pregnancy test. To take part in this study, you must not be pregnant.

A series of tests used to check your nerve function will also be performed. In total, it should take about 1-2 hours to complete these 4 tests. The following nerve function tests will be performed:

* You will complete hand tasks, such as writing, card turning, picking up small objects, and stacking). You will also be timed as you insert 25 shaped pegs into a board.
* You will complete 2 balance tests. The first balance test measures how long you can stand on 1 leg. The second balance test measures your ability to stand up from a chair, walk about 10 feet, and return back to the chair.

Acupuncture Sessions:

At each session, before you receive the acupuncture, your tongue checked and your heart rate will be measured.

Your first acupuncture session may be on the same day as some of the tests described above, if possible. If not, it will be scheduled for another day no more than 14 days after the screening visit, unless you are in Group 3.

For each session, you will be placed in a comfortable position and the study doctor/acupuncturist will find points on your body where the needles will be placed. All study participants will have the needles placed at the same points on the body (the hands, feet, legs, abdomen, and scalp).

Very thin, solid, sterile, stainless steel needles will be used. All of the needles are specially made for acupuncture. The depth of the needle in the skin and the number of needles used is based on standard acupuncture procedures. The needles will remain in place for about 20 minutes.

Electrical stimulation will be added to some of the needles on your feet and hands. This involves placing wires on the needles, which are connected to a machine that delivers a weak electrical current through the wires. The strength of the electrical current will be changed slowly until it is at a comfortable level for you.

Most acupuncture sessions will last about 1 hour. On the weeks that you complete the questionnaires, it will add about 15-20 minutes.

After your 6th and 12th acupuncture sessions, you will complete the same 3 questionnaires as you did at the beginning of the study.

Length of Study:

You may take part in this study for up to 28 weeks. If intolerable side effects or symptoms occur, you will be taken off study early.

End-of-Study Visit:

At the end of the study, or if you go off study early for any reason, you will have an end-of-study visit. If the doctor thinks it is needed, the following procedures will be performed within 4 weeks after your last acupuncture session:

* You will complete the same 3 questionnaires as before.
* The 4 nerve tests will be repeated in order to learn if there have been any changes in your nerve function.
* Your tongue will be checked and your heart rate will be measured.

Additional Information:

During the study, you may still receive your regular pain treatments. You should tell the study doctor if you want to change your dose or want to start any new drugs for the treatment of your neuropathy.

If you were in Group 2 or 3, after your participation on this study is complete, you may receive 3 extra acupuncture treatments.

This is an investigational study. The acupuncture needles used in this study are commercially available and FDA approved. It is considered investigational to use acupuncture to treat peripheral neuropathy related to chemotherapy.

Up to 120 patients will take part in this multicenter study. Up to 60 will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have the ability to understand English, Mandarin, or Taiwanese.
2. Sign a written informed consent document.
3. Willing to follow protocol requirements.
4. Age 18 and older.
5. History of diagnosis of cancer.
6. Patients must have neuropathy greater or equal to 2 according to CTCAE v 4.0 scale despite previous treatment, which may include Neurontin, Cymbalta and/or Lyrica. Patients receiving any of these drugs must remain on the same medications throughout the study period; however, adjustments in dosage are allowed. Patients will be removed from the study if a change in type of medication is necessary. Patients are allowed to stop medications but not replace them with other medications
7. The patient's previous chemotherapy treatment must have included a taxane (paclitaxel, nab-paclitaxel, or docetaxel) or platinum (cisplatin, oxaliplatin, or carboplatin) and considered the primary cause of the neuropathy by the medical team.
8. ECOG Performance Status of 0, 1, or 2 (Appendix B).
9. Willingness to comply with all study interventions of acupuncture and follow-up assessments.

Exclusion Criteria:

1. Current active treatment with chemotherapy, radiation or surgery in the past 3 months or planned treatment during this study protocol period. Hormonal therapy is allowed.
2. Treatment with any neuropathic agent including taxane, platinum, vinca alkaloid, or bortezumab chemotherapy in the past 6 months.
3. Local infection at or near the acupuncture site. (Although acupuncture is a minimally invasive procedure, patients will be excluded if there is an indication of infection.)
4. Physical deformities that could interfere with accurate acupuncture point location.
5. Concurrent use of other alternative medicines such as herbal agents and high dose vitamins and minerals.
6. Known coagulopathy or taking heparin (including low molecular weight heparin) at full anti-coagulation doses (prophylaxis is allowed) or Coumadin at any dose. Patients on aspirin or non-steroidal anti-inflammatories or other antiplatelet medicines will be allowed to participate.
7. Platelets < 50 H K/UL in the past 30 days.
8. WBCs < 3.0 K/UL or ANC <1,500 K/UL) in the past 30 days.
9. Active CNS disease. (The action for acupuncture may be associated with central nervous system activity, and patients with CNS pathology may respond differently to treatment than the general population.)
10. Cardiac pacemaker.
11. Mental incapacitation or significant emotional or psychological disorder that, in the opinion of the investigators, precludes study entry. (These patients may not be able to cooperate with this slightly invasive procedure or with the data collection process.)
12. Currently pregnant. (Certain acupuncture applications have been reported to stimulate uterine contractions.)
13. History of diabetic neuropathy or neuropathy related to HIV.
14. Previous acupuncture treatment for any indication within 30 days of enrollment.
15. Planned or actual changes in type of medications that could affect symptoms related to PN. New medications for the treatment of CIPN are not allowed during the study. Note: Subjects need to be on stable doses of CIPN medications for 4 weeks.
16. Grade III lymphedema or lymphedema considered severe by the treating clinician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Acupuncture With or Without Electrical Stimulation | After 24 acupuncture treatments
  Difference in scores compared from baseline to 24 treatments between the two groups with or without electrical stimulations using two-sample t-test. Difference between baseline and 24 treatments assessed in the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group (FACT/GOG)-Neurotoxicity (Ntx) subscale scores separately for each of the 2 acupuncture schedules using a paired t test.
Difference in Acupuncture Response | After 12 and 24 acupuncture treatments
  Effect of 12 versus 24 acupuncture treatments examined for symptoms of chronic, chemotherapy-induced peripheral neuropathy in cancer patients and survivors. Efficacy analysis estimated using average difference between 12-week assessment and 24-week assessment in the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group (FACT/GOG)-Neurotoxicity (Ntx) scale for each acupuncture schedule using a paired t test. Response difference examined between 12 versus 24 acupuncture treatments using analysis of variance including the two treatment schedules and the indicator of receiving electrical stimulation as the factors, and considering the interaction between the two factors.

SECONDARY OUTCOMES:
Comparison of Symptom Scores | 14 weeks after randomization
  Symptom scores of the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group (FACT/GOG)-Neurotoxicity (Ntx) scale compared between the waitlist control and the acupuncture treatment groups at week 14 after randomization compared using two-sample t-test or Wilcoxon rank-sum test.

CONTACTS AND LOCATIONS:
Overall Officials: Richard T. Lee, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org